CLINICAL TRIAL: NCT01782859
Title: Effect of Steroids Given Over 24 Hours on Cytokine Release, Urinary Desmosine Level and Thrombogenic Markers in Patients Undergoing Unilateral Total Hip Replacement
Brief Title: Effect of Steroids on Thrombosis (Blood Clot Formation) and Inflammation in Patients Undergoing Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-008
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Results first posted 2016-05-10 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-07

CONDITIONS: Total Hip Replacement
MeSH Terms: interventions — Prednisone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Control group
  Interventions: Drug: Placebo (for Prednisone)
- Prednisone/hydrocortisone (Active Comparator): Steroid group will receive the following:
  1. 20 mg prednisone pill to be taken in the morning of surgery prior to arrival to the hospital
  2. 100 mg hydrocortisone IV 8 hours after first dose of prednisone followed by 3. Second and last dose of 100 mg hydrocortisone IV
  Interventions: Drug: Prednisone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Prednisone
  Other Names: Low dose steroids to be administered preoperatively and then repeated over a 24-hour period; 1. 20 mg prednisone pill to be taken in the morning of surgery prior to arrival to the hospital; 2. 100 mg hydrocortisone IV 8 hours after first dose of prednisone followed by; 3. Another dose of 100 mg hydrocortisone IV 8 hours after
  Arms: Prednisone/hydrocortisone
Drug: Hydrocortisone
  Other Names: Low dose steroids to be administered preoperatively and then repeated over a 24-hour period; 1. 20 mg prednisone pill to be taken in the morning of surgery prior to arrival to the hospital; 2. 100 mg hydrocortisone IV 8 hours after first dose of prednisone followed by; 3. Another dose of 100 mg hydrocortisone IV 8 hours after
  Arms: Prednisone/hydrocortisone
Drug: Placebo (for Prednisone)
  Other Names: Lactose filler to mimic 20 mg prednisone tablet
  Arms: Placebo

SUMMARY:
Studies have shown that surgery causes some reactions in your body consistent with inflammation. When the inflammation is extensive, it may affect different parts of the body including the lungs. Corticosteroids are commonly used to treat inflammation and are different from performance enhancing steroids associated with athletics. The purpose of this study is to determine the influence of low dose steroids given 3 times in a 24 hour period on thrombotic markers (markers that are associated with increased risks of clotting, a possible complication of surgery), interleukin (IL)-6 cytokine release (part of the stress response seen with surgery), and urine desmosine levels (a marker of lung injury) in a randomized placebo controlled trial patients undergoing total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total hip replacement with Drs. Douglas Padgett, Thomas Sculco, or Edwin Su.
* Patients between the age of 50 and 90

Exclusion Criteria:

* Patients on steroid therapy regardless of dose or duration of treatment or those requiring stress-dose steroids preoperatively
* Patients who are smokers
* Patients who have diabetes
* Patients who are <50 and >90 years of age
* Patients with history of prior difficulties tolerating corticosteroids

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Control group
  Placebo (for Prednisone)
Period: Overall Study
Arm/Group | Placebo | Prednisone/Hydrocortisone
Started | 20 | 20
Completed | 14 | 13
Not Completed | 6 | 7
Not completed — Protocol Violation | 6 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Prednisone/Hydrocortisone | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.13 (7.16) | 66.21 (8.80) | 65.66 (7.87)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Body mass index [Mean (Standard Deviation); unit: kg/(m^2)] | 26.04 (3.92) | 28.03 (4.86) | 27.00 (4.43)

OUTCOME MEASURES:

1. Primary Outcome: Serum Prothrombin Fragment 1 and 2 (PF 1.2)
Time Frame: First 24 hours after surgery
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | Prednisone/Hydrocortisone
Number analyzed (Participants) | 14 | 13
pmol/mL
  Baseline | 334.15 (193.9) | 298.12 (124.6)
  Wound Closure | 778.33 (353.7) | 619.21 (154.9)
  4 hours postoperatively | 1306.76 (445.4) | 1138.65 (435.7)
  6 hours postoperatively | 1175.71 (400.9) | 1032.52 (466.8)
  24 hours postoperatively | 356.79 (94.9) | 422.61 (191.6)

2. Primary Outcome: Plasmin-a 2 Antiplasmin Complex (PAP)
Time Frame: First 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | Prednisone/Hydrocortisone
Number analyzed (Participants) | 14 | 13
mcg/L
  Baseline | 924.67 (324.7) | 1011.17 (212.3)
  Wound Closure | 1361.23 (527.7) | 2251.33 (680.1)
  4 hours postoperatively | 2251.33 (680.1) | 2455.71 (458.0)
  6 hours postoperatively | 2283.18 (711.0) | 2379.57 (395.3)
  24 hours postoperatively | 996.39 (251.1) | 914.16 (186.6)

3. Secondary Outcome: Interleukin (IL)-6 Cytokine Release (Inflammatory Marker)
Description: The time frame of the study for each patient covers the period between time of surgery and until discharge from the hospital.
Time Frame: Participants will be followed from the time of surgery until discharge, expected average of 3-5 days
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Placebo | Prednisone/Hydrocortisone
Number analyzed (Participants) | 14 | 13
picograms/milliliter
  Baseline | 2.98 (2.3) | 5.69 (8.7)
  Wound closure | 4.46 (4.2) | 4.47 (6.3)
  4 hours postoperatively | 89.21 (52.1) | 56.72 (27.6)
  6 hours postoperatively | 115.17 (56.1) | 64.4 (33.7)
  24 hours postoperatively | 176.79 (91.4) | 68.51 (45.8)

4. Secondary Outcome: Desmosine Level (Marker of Lung Injury)
Description: as for outcome 3
Time Frame: Participants will be followed from the time of surgery until discharge, expected average of 3-5 days
Population: Desmosine levels were not analyzed.
Arm/Group | Placebo | Prednisone/Hydrocortisone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain at 3 Months Post-op
Description: At 3 months postoperatively, patients were asked to rate their pain on a scale of 0-10, with 0 being no pain and 10 being worst pain.
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prednisone/Hydrocortisone: Steroid group will receive the following:
  1. 20 mg prednisone pill to be taken in the morning of surgery prior to arrival to the hospital
  2. 100 mg hydrocortisone IV 8 hours after first dose of prednisone followed by 3. Second and last dose of 100 mg hydrocortisone IV
  Prednisone
  Hydrocortisone
Arm/Group | Placebo | Prednisone/Hydrocortisone
Number analyzed (Participants) | 14 | 13
units on a scale | 0.92 (0.76) | 0.54 (0.66)

ADVERSE EVENTS:
Arm/Group | Placebo | Prednisone/Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes